CLINICAL TRIAL: NCT05450328
Title: Inhaled Milrinone and Epoprostenol for the Prevention of Difficult Cardiac Pulmonary Bypass Separation: A Randomized, Double-blind, Controlled Trial
Brief Title: Inhaled Milrinone and Epoprostenol for the Prevention of Difficult Cardiac Pulmonary Bypass Separation
Acronym: MILAN
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ICM 2022-3026
Record Dates: First submitted 2022-05-16; First posted 2022-07-08 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Right Heart Failure; Right Ventricular Dysfunction
Keywords: Cardiac Surgery; Right Ventricular Dysfunction; Cardiopulmonary Bypass; Inhaled Therapy
MeSH Terms: conditions — Heart Failure; Ventricular Dysfunction, Right | interventions — Milrinone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Normal Saline (Placebo Comparator): The control group will receive a saline solution (8mL) as a placebo, before CPB start.
  Interventions: Drug: Normal saline
- Combination of inhaled Epoprostenol and Milrinone (Active Comparator): The experimental group will receive simultaneously 4mg of Milrinone (1mg/mL, 4mL) and 60 mcg of Epoprostenol (15 mcg/mL, 4mL) before CPB initiation.
  Interventions: Drug: Combined Epoprostenol Sodium & Milrinone

INTERVENTIONS:
Drug: Combined Epoprostenol Sodium & Milrinone — One syringe containing 4mg of milrinone (1mg/mL, 4mL) and one syringe containing 60 mcg of epoprostenol (15 mcg/mL, 4mL).
  The drugs will be administered via an ultrasonic nebulizer (Aeroneb Professional Nebulizer System, Aerogen Ltd, Galway, Ireland, registration number: 66728) over a period of 20 minutes. This type of nebulizer is used routinely at the Montreal Heart Institute and can hold a maximum of 8 mL of solutions.
  Arms: Combination of inhaled Epoprostenol and Milrinone
Drug: Normal saline — The control group will receive two syringes of 4mL of Normal Saline, before CPB start.
  The placebo will be administered via an ultrasonic nebulizer (Aeroneb Professional Nebulizer System, Aerogen Ltd, Galway, Ireland, registration number: 66728) over a period of 20 minutes. This type of nebulizer is used routinely at the Montreal Heart Institute and can hold a maximum of 8 mL of solutions.
  Arms: Normal Saline

SUMMARY:
In cardiac surgery, the presence of pulmonary hypertension (PH) is a prognostic factor associated with increased mortality and morbidity. In this context, one of the main causes of PH is related to reperfusion ischemia during weaning from extracorporeal circulation (CPB). One of the consequences of PH is right ventricular dysfunction. During weaning from CPB, the development of a right ventricular dysfunction is associated with increased requirements for vasopressor and inotropic agents, duration of mechanical ventilation, prolonged intensive care and hospital stay, and increased mortality compared with patients with left ventricular (LV) dysfunction. The management of patients with PH with or without right ventricular (RV) dysfunction relies on several strategies such as the administration of intravenous and inhaled agents, or mechanical ventricular support. Among those agents, the administration of inotropes or pulmonary vasodilators such as epoprostenol, milrinone and nitric oxide are among the most widely used treatments recommended by the Canadian Cardiovascular Society. At the Montreal Heart Institute, inhaled epoprostenol and milrinone are routinely administered to patients with PH or LV dysfunction in the perioperative setting. Despite the frequent use of inhaled epoprostenol and milrinone, Health Canada has not yet approved the use of these molecules.

The primary objective of this multicenter, double-blind, randomized clinical trial is to evaluate the clinical efficacy of the combined administration of inhaled epoprostenol and milrinone in a cardiac surgery setting. This trial will compare the clinical outcome of 71 patients who will receive inhaled epoprostenol and milrinone before the start of bypass surgery to 71 patients who will receive a placebo before the start of the CPB. The primary clinical outcome is the proportion of patients with an "unsuccessful" CPB weaning defined by the use of an inotrope +/- vasopressor agent or the use of mechanical circulatory support or a return to bypass grafting for hemodynamic reasons.

This clinical trial will evaluate the clinical efficacy of the combination of inhaled agents in a cardiac surgery setting. Therefore, if the results of this study are positive, the combination of inhaled epoprostenol and milrinone will optimize the management of patients with pulmonary hypertension with or without a right ventricular dysfunction.

DETAILED DESCRIPTION:
Hypothesis: Based on the knowledge gained from previous work, the administration of inhaled Milrinone and Epoprostenol therapy prior to the initiation of cardiopulmonary bypass (CPB) is superior in terms of favourable clinical outcomes. The combined administration of these agents improves right ventricular performance while reducing myocardial and pulmonary ischemia-reperfusion injury secondary to weaning from bypass surgery. For these reasons, we hypothesize that administration of combination therapy before the start of CPB may provide better hemodynamic stability throughout the surgery and favourable postoperative clinical outcomes.

Objective:

Primary Objective To determine whether the use of inhaled Epoprostenol and Milrinone, prior to the initiation of CPB, decreases the occurrence of difficult CPB weaning compared to placebo administration.

Secondary Objectives To determine the effect of combined use of inhaled Epoprostenol and Milrinone, prior to the initiation of CPB on hemodynamic and perioperative parameters.

To determine the effect of combined use of inhaled Epoprostenol and milrinone, prior to the initiation of CPB on postoperative clinical outcomes.

Design: The proposed study is a randomized, double-blind, controlled trial to determine the efficacy of the combined use of inhaled Epoprostenol and Milrinone prior to the initiation of CPB compared with the use of a placebo in a cardiac surgery setting. The clinical outcome of interest is the incidence of a difficult weaning from CPB. A difficult weaning is defined as the use of an inotrope with or without a vasopressor agent or the use of mechanical circulatory support or a return on CPB for hemodynamic reasons.

Patients/Participants:

Inclusion Criteria Only patients undergoing cardiac surgery with CPB and aged 18 years and older will be included in this study.

Interventions:

We will randomly assign the 142 patients in a 1:1 allocation scheme to receive a combination of inhaled Epoprostenol and Milrinone or a placebo after induction of general anesthesia, i.e. before CPB initiation. Free and informed consent to participate in this research project will be obtained the day before surgery by the anesthesiologist in charge of the case or by a member of the research team.

In both study groups, the anesthetic procedure will be performed according to Canadian practice standards and is left to the discretion of the clinician. In both groups, the procedure will be administered via an ultrasonic nebulizer (Aeroneb Professional Nebulizer System, Aerogen Ltd, Galway, Ireland, registration number: 66728) over a period of 20 minutes. This type of nebulizer is used routinely at the Montreal Heart Institute and can hold a maximum of 8 mL of solutions.

The experimental group will receive simultaneously 4mg of Milrinone (1mg/mL, 4mL) and 60 mcg of Epoprostenol (15 mcg/mL, 4mL) before CPB initiation. The control group will receive a saline solution (8mL) as a placebo, before CPB start. For each patient, 2 syringes of 4mL will be prepared on the morning of surgery, depending on the allocation group, to ensure drug stability. For example, for patients in the experimental group, one syringe containing 4mg of milrinone (1mg/mL, 4mL) and one syringe containing 60 mcg of epoprostenol (15 mcg/mL, 4mL) will be prepared. For the control group, two syringes containing 4mL of 0.9% physiological saline will be prepared.

Expected outcomes:

The administration of this combination therapy prior to the start CPB may decrease the proportion of patients presenting a difficult CPB weaning, in addition to better hemodynamic stability during surgery. Also, we believe that patients who have received the combined therapy will have favourable postoperative clinical outcomes, such as less vasoactive and inotropic agents and a reduction in the duration of postoperative organ dysfunction.

This randomized, double-blind, multicenter, controlled clinical trial will evaluate the clinical efficacy of the combination of inhaled agents in cardiac surgery setting intraoperatively and postoperatively. Therefore, if the results of this study are positive, the combination of inhaled Epoprostenol and Milrinone will optimize the management of patients with pulmonary hypertension with or without right ventricular dysfunction.

ELIGIBILITY:
Inclusion Criteria:

- Only patients undergoing cardiac surgery with CPB and aged 18 years and older will be included in this study.

Exclusion Criteria:

* The presence of congenital cardiomyopathy, which the correction is the primary objective of the proposed surgery. For example, a patient who requires surgery for atrial septal defect closure only would not be eligible for the study. On the other hand, a patient who undergoes this same surgery in addition to a valve replacement, for example, would be eligible to participate in the study.
* Heart transplant or ventricular assist device surgery
* Urgent surgery including hemodynamic instability requiring vasopressor agents upon arrival in the operating room
* A contraindication to transesophageal ultrasound monitoring or the presence of an unstable cervical spine.
* Presence of a contraindication related to Epoprostenol or Milrinone administration such as a documented left ventricular or right ventricular outflow tract obstruction, a severe unaddressed aortic stenosis, or a documented allergy to either of these two molecules.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 141 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who have a difficult CPB weaning in both groups | 1 year
  To determine whether the use of inhaled Epoprostenol and Milrinone, prior to the initiation of CPB, decreases the occurrence of difficult CPB weaning compared to placebo administration.

SECONDARY OUTCOMES:
Correlation between the variation of central venous pressure and patients who received the treatment | 1 year
  To determine the effect of combined use of inhaled Epoprostenol and Milrinone, prior to the initiation of CPB on central venous pressure.
Correlation between the variation of cardiac output and patients who received the treatment | 1 year
  To determine the effect of combined use of inhaled Epoprostenol and milrinone, prior to the initiation of CPB on cardiac output.
Correlation between the variation of arterial pressure and patients who received the treatment | 1 year
  To determine the effect of combined use of inhaled Epoprostenol and milrinone, prior to the initiation of CPB on arterial pressure.
Correlation between the right ventricular curve etiology (normal, square root, oblique) and patients who received the treatment | 1 year
  To determine the effect of combined use of inhaled Epoprostenol and milrinone, prior to the initiation of CPB on right ventricular curve etiology.
Correlation between the PAM/ PAPM ratio taken at T0 and T1 and patients who received the treatment | 1 year
  To determine the effect of combined use of inhaled Epoprostenol and milrinone, prior to the initiation of CPB on PAM/PAPM ratio.
Correlation between the cardiac index taken at T0 and T1 and patients who received the treatment | 1 year
  To determine the effect of combined use of inhaled Epoprostenol and milrinone, prior to the initiation of CPB on cardiac index.
Correlation between right ventricular contractility and patients who received the treatment | 1 year
  To determine the effect of combined use of inhaled Epoprostenol and milrinone, prior to the initiation of CPB on the dp/dt calculated from the right ventricular waveform.
Correlation between right ventricular outflow tract obstruction and patients who received the treatment | 1 year
  To determine the effect of combined use of inhaled Epoprostenol and milrinone, prior to the initiation of CPB on right ventricular systolic pressure and systolic pulmonary artery pressure variation.
Correlation between cerebral saturation and patients who received the treatment | 1 year
  To determine the effect of combined use of inhaled Epoprostenol and milrinone, prior to the initiation of CPB on the cerebral saturation quantified by the near infrared spectroscopy.
Correlation between fluid administration during surgery and patients who received the treatment | 1 year
  To determine the effect of combined use of inhaled Epoprostenol and milrinone, prior to the initiation of CPB on fluid administration during surgery such as crystalloid, colloid and blood transfusion.
Correlation between the vasoactive and inotropic score and patients who received the treatment | 1 year
  To determine the effect of combined use of inhaled Epoprostenol and milrinone, prior to the initiation of CPB on the vasoactive and inotropic score quantified on the patient arrival in the ICU.
Correlation between the time of persistent organ dysfunction (TPOD) and patients who received the treatment | 1 year
  To determine the effect of combined use of inhaled Epoprostenol and milrinone, prior to the initiation of CPB on the TPOD.
Correlation between the ICU stay and patients who received the treatment | 1 year
  To determine the effect of combined use of inhaled Epoprostenol and milrinone, prior to the initiation of CPB on the ICU stay.
Correlation between the post-operative complications and patients who received the treatment | 1 year
  To determine the effect of combined use of inhaled Epoprostenol and milrinone, prior to the initiation of CPB on post-operative complications defined by the Society of Thoracic Surgeons and patients who received the treatment.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Denault AY, Bussieres JS, Arellano R, Finegan B, Gavra P, Haddad F, Nguyen AQN, Varin F, Fortier A, Levesque S, Shi Y, Elmi-Sarabi M, Tardif JC, Perrault LP, Lambert J. A multicentre randomized-controlled trial of inhaled milrinone in high-risk cardiac surgical patients. Can J Anaesth. 2016 Oct;63(10):1140-1153. doi: 10.1007/s12630-016-0709-8. Epub 2016 Jul 28. PMID 27470232
- [Result] Davila-Roman VG, Waggoner AD, Hopkins WE, Barzilai B. Right ventricular dysfunction in low output syndrome after cardiac operations: assessment by transesophageal echocardiography. Ann Thorac Surg. 1995 Oct;60(4):1081-6. doi: 10.1016/0003-4975(95)00526-q. PMID 7574953
- [Result] Authors/Task Force Members; Kunst G, Milojevic M, Boer C, De Somer FMJJ, Gudbjartsson T, van den Goor J, Jones TJ, Lomivorotov V, Merkle F, Ranucci M, Puis L, Wahba A; EACTS/EACTA/EBCP Committee Reviewers; Alston P, Fitzgerald D, Nikolic A, Onorati F, Rasmussen BS, Svenmarker S. 2019 EACTS/EACTA/EBCP guidelines on cardiopulmonary bypass in adult cardiac surgery. Br J Anaesth. 2019 Dec;123(6):713-757. doi: 10.1016/j.bja.2019.09.012. Epub 2019 Oct 2. No abstract available. PMID 31585674
- [Result] El Kebir D, Hubert B, Taha R, Troncy E, Wang T, Gauvin D, Gangal M, Blaise G. Effects of inhaled nitric oxide on inflammation and apoptosis after cardiopulmonary bypass. Chest. 2005 Oct;128(4):2910-7. doi: 10.1378/chest.128.4.2910. PMID 16236968
- [Result] McMullan DM, Bekker JM, Parry AJ, Johengen MJ, Kon A, Heidersbach RS, Black SM, Fineman JR. Alterations in endogenous nitric oxide production after cardiopulmonary bypass in lambs with normal and increased pulmonary blood flow. Circulation. 2000 Nov 7;102(19 Suppl 3):III172-8. doi: 10.1161/01.cir.102.suppl_3.iii-172. PMID 11082382
- [Result] Seghaye MC, Duchateau J, Bruniaux J, Demontoux S, Detruit H, Bosson C, Lecronier G, Mokhfi E, Serraf A, Planche C. Endogenous nitric oxide production and atrial natriuretic peptide biological activity in infants undergoing cardiac operations. Crit Care Med. 1997 Jun;25(6):1063-70. doi: 10.1097/00003246-199706000-00026. PMID 9201062
- [Result] Lamarche Y, Malo O, Thorin E, Denault A, Carrier M, Roy J, Perrault LP. Inhaled but not intravenous milrinone prevents pulmonary endothelial dysfunction after cardiopulmonary bypass. J Thorac Cardiovasc Surg. 2005 Jul;130(1):83-92. doi: 10.1016/j.jtcvs.2004.09.011. PMID 15999045
- [Result] Lamarche Y, Perrault LP, Maltais S, Tetreault K, Lambert J, Denault AY. Preliminary experience with inhaled milrinone in cardiac surgery. Eur J Cardiothorac Surg. 2007 Jun;31(6):1081-7. doi: 10.1016/j.ejcts.2007.02.019. Epub 2007 Apr 2. PMID 17400468
- [Result] Haddad F, Denault AY, Couture P, Cartier R, Pellerin M, Levesque S, Lambert J, Tardif JC. Right ventricular myocardial performance index predicts perioperative mortality or circulatory failure in high-risk valvular surgery. J Am Soc Echocardiogr. 2007 Sep;20(9):1065-72. doi: 10.1016/j.echo.2007.02.017. Epub 2007 Jun 12. PMID 17566702
- [Result] Maslow AD, Regan MM, Panzica P, Heindel S, Mashikian J, Comunale ME. Precardiopulmonary bypass right ventricular function is associated with poor outcome after coronary artery bypass grafting in patients with severe left ventricular systolic dysfunction. Anesth Analg. 2002 Dec;95(6):1507-18, table of contents. doi: 10.1097/00000539-200212000-00009. PMID 12456409
- [Result] Haddad F, Doyle R, Murphy DJ, Hunt SA. Right ventricular function in cardiovascular disease, part II: pathophysiology, clinical importance, and management of right ventricular failure. Circulation. 2008 Apr 1;117(13):1717-31. doi: 10.1161/CIRCULATIONAHA.107.653584. No abstract available. PMID 18378625
- [Result] Denault AY, Tardif JC, Mazer CD, Lambert J; BART Investigators. Difficult and complex separation from cardiopulmonary bypass in high-risk cardiac surgical patients: a multicenter study. J Cardiothorac Vasc Anesth. 2012 Aug;26(4):608-16. doi: 10.1053/j.jvca.2012.03.031. Epub 2012 May 11. PMID 22578975
- [Result] Hirani N, Brunner NW, Kapasi A, Chandy G, Rudski L, Paterson I, Langleben D, Mehta S, Mielniczuk L; CCS/CTS Pulmonary Hypertension Committee. Canadian Cardiovascular Society/Canadian Thoracic Society Position Statement on Pulmonary Hypertension. Can J Cardiol. 2020 Jul;36(7):977-992. doi: 10.1016/j.cjca.2019.11.041. PMID 32682511
- [Result] Haj RM, Cinco JE, Mazer CD. Treatment of pulmonary hypertension with selective pulmonary vasodilators. Curr Opin Anaesthesiol. 2006 Feb;19(1):88-95. doi: 10.1097/01.aco.0000192765.27453.5a. PMID 16547439
- [Result] Elmi-Sarabi M, Deschamps A, Delisle S, Ased H, Haddad F, Lamarche Y, Perrault LP, Lambert J, Turgeon AF, Denault AY. Aerosolized Vasodilators for the Treatment of Pulmonary Hypertension in Cardiac Surgical Patients: A Systematic Review and Meta-analysis. Anesth Analg. 2017 Aug;125(2):393-402. doi: 10.1213/ANE.0000000000002138. PMID 28598920
- [Result] Green JB, Hart B, Cornett EM, Kaye AD, Salehi A, Fox CJ. Pulmonary Vasodilators and Anesthesia Considerations. Anesthesiol Clin. 2017 Jun;35(2):221-232. doi: 10.1016/j.anclin.2017.01.008. Epub 2017 Apr 14. PMID 28526144
- [Result] Fox BD, Shtraichman O, Langleben D, Shimony A, Kramer MR. Combination Therapy for Pulmonary Arterial Hypertension: A Systematic Review and Meta-analysis. Can J Cardiol. 2016 Dec;32(12):1520-1530. doi: 10.1016/j.cjca.2016.03.004. Epub 2016 Mar 17. PMID 27378592
- [Result] Hache M, Denault AY, Belisle S, Couture P, Babin D, Tetrault F, Guimond JG. Inhaled prostacyclin (PGI2) is an effective addition to the treatment of pulmonary hypertension and hypoxia in the operating room and intensive care unit. Can J Anaesth. 2001 Oct;48(9):924-9. doi: 10.1007/BF03017361. PMID 11606352
- [Result] Hardy JF, Belisle S. Inotropic support of the heart that fails to successfully wean from cardiopulmonary bypass: the Montreal Heart Institute experience. J Cardiothorac Vasc Anesth. 1993 Aug;7(4 Suppl 2):33-9. doi: 10.1016/1053-0770(93)90095-3. PMID 8103681
- [Result] Blaise G, Langleben D, Hubert B. Pulmonary arterial hypertension: pathophysiology and anesthetic approach. Anesthesiology. 2003 Dec;99(6):1415-32. doi: 10.1097/00000542-200312000-00027. No abstract available. PMID 14639158
- [Result] Gaies MG, Gurney JG, Yen AH, Napoli ML, Gajarski RJ, Ohye RG, Charpie JR, Hirsch JC. Vasoactive-inotropic score as a predictor of morbidity and mortality in infants after cardiopulmonary bypass. Pediatr Crit Care Med. 2010 Mar;11(2):234-8. doi: 10.1097/PCC.0b013e3181b806fc. PMID 19794327
- [Result] Shahian DM, O'Brien SM, Filardo G, Ferraris VA, Haan CK, Rich JB, Normand SL, DeLong ER, Shewan CM, Dokholyan RS, Peterson ED, Edwards FH, Anderson RP; Society of Thoracic Surgeons Quality Measurement Task Force. The Society of Thoracic Surgeons 2008 cardiac surgery risk models: part 1--coronary artery bypass grafting surgery. Ann Thorac Surg. 2009 Jul;88(1 Suppl):S2-22. doi: 10.1016/j.athoracsur.2009.05.053. PMID 19559822
- [Result] van Heerden PV, Gibbs NM, Michalopoulos N. Effect of low concentrations of prostacyclin on platelet function in vitro. Anaesth Intensive Care. 1997 Aug;25(4):343-6. doi: 10.1177/0310057X9702500402. PMID 9288373